CLINICAL TRIAL: NCT03695588
Title: Quadratus Lumborum Block (QLB) for Pain Relief After Caesarean Section: A Prospective, Double-blind, Randomised Controlled Trial.
Brief Title: Quadratus Lumborum Block (QLB) for Pain Relief After Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coombe Women and Infants University Hospital (Other)
Responsible Party: Principal Investigator, Ruairi Irwin, Principal investigator, Coombe Women and Infants University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CWIUH-QLB
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Quadratus Lumborum Block
Keywords: pain relief; Caesarean; Cesarean; c-section; intrathecal morphine; analgesia; QLB; QL; QLB2; QL2
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum block (Active Comparator): Bilateral posterior QLB with 20ml 0.25% L-Bupivacaine.
  Interventions: Procedure: Quadratus lumborum block
- Sham QLB (Sham Comparator): Sham QLB - Ultrasound identification of QLB followed by skin pressure with blunt needle. Patient blinded due to residual spinal anaesthetic block.
  Interventions: Procedure: Sham QLB

INTERVENTIONS:
Procedure: Quadratus lumborum block — Ultrasound guided Quadratus Lumborum block using a posterior approach. (QLB 2)
  Arms: Quadratus lumborum block
Procedure: Sham QLB — Sham QLB - Ultrasound identification of QLB followed by skin pressure with blunt needle.
  Arms: Sham QLB

SUMMARY:
There is currently a gap in the literature with regards to the utility of the QLB performed in conjunction with intrathecal morphine (ITM) for Caesarean section. The aim of the study is to assess the efficacy of the QLB as part of a multi-modal analgesic approach in patients after caesarean section.

DETAILED DESCRIPTION:
Post-operative pain relief management remains challenging after Caesarean-section. The perfect postoperative analgesic regimen is yet to be elucidated, but opioids remain a cornerstone whether they are administered intra-thecally, or systemically or both. Unfortunately, opioids are associated with significant adverse effects such as respiratory depression, post-operative nausea and vomiting (PONV), sedation and pruritus. Therefore, the search for opioid sparing analgesic techniques is important.

The study treatment consists of a quadratus lumborum block (QLB) of either 0.25% Levobupivacaine or a simulated sham QLB after C-section under spinal anaesthesia. The participants will be randomized into one of two groups with an internet based randomisation tool, and then allocated to either group as per the allocation in a sealed opaque envelope.

Spinal anaesthesia will be performed in a standardised manner using 10-15mg hyperbaric bupivacaine, 20ug fentanyl and 100ug preservative free morphine. Anaesthetic and surgical management will be conducted as per the usual manner. Diclofenac 100mg suppositories and IV Paracetamol 1g will be administered at the end of surgery. A Morphine PCA will be connected to the patient in the recovery room after the intervention.

The bilateral posterior QLB will be performed after surgery in the supine position in an aseptic manner. The patient will be blinded to the group intervention as the sterile drapes will be left hanging blocking the patient's view of the procedure. The block from the spinal anaesthetic will mean the patient is unaware of the procedure being carried out. A curvilinear ultrasound probe will be used to identify the quadratus lumborum muscle.

Intervention group:

Aseptic, ultrasound guided, bilateral QLB using a posterior approach. This is known as the QLB 2 approach. A maximum volume of 20 ml of 0.25% Levobupivacaine will be administered each side. After the procedure a sterile dressing will be placed on the puncture site.

Placebo group:

The patient will be sterilized, draped and scanned in the same manner as the intervention group, until the target injection point is identified. The operator will use a blunt needle to apply pressure to the skin, (without breaking the skin), for one minute as if they are performing the procedure. This will be performed bilaterally. After the procedure, a sterile dressing will be placed over the pressure area.

ELIGIBILITY:
Inclusion Criteria:

* Elective Caesarean section under spinal anaesthesia.
* Age > 18 years old.
* Singleton pregnancy.

Exclusion Criteria:

* Contraindication to spinal or regional anaesthesia.
* Allergy/sensitivity/contraindication to study medications.
* Unable to comprehend visual analogue scale.
* BMI > 40.
* Booking weight <40kg.
* History of chronic pain or regular opioid use.
* Pre-eclampsia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
IV PCA Morphine consumption up to 24 hours. | 24 hours
  Intravenous PCA (patient controlled analgesia) morphine consumption up to 24 hours.

SECONDARY OUTCOMES:
Pain scores at rest. | 6, 12, 24, 48 hours
  VAS (visual analogue scale) pain scores at rest - lying supine in bed.
Pain scores on movement. | 6, 12, 24, 48 hours
  VAS pain scores on movement - raising head and shoulders off pillow when lying supine in bed.
Nausea and vomiting. | 24, 48 hours
  The incidence of N+V requiring rescue anti-emetics.
IV PCA morphine bolus demands. | 24 hours
  Intravenous PCA (patient controlled analgesia) morphine bolus demands up to 24 hours.
Total opioid consumption at 48 hours. | 48 hours
  Total opioid consumption at 48 hours - converted to IV morphine equivalents.
QbsQoR-11. | 24, 48 hours
  Quality of Recovery questionnaire.
QoR-15. | 24, 48 hours
  Quality of Recovery questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Tan, Principal Investigator — Head of Department of Anaesthesia CWIUH
Locations (1):
- Coombe Women and Infants University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No